CLINICAL TRIAL: NCT03790800
Title: Intensive Ambulance-delivered Blood Pressure Reduction in Hyper-Acute Stroke Trial
Acronym: INTERACT4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Shanghai East Hospital, China (Unknown); First Affiliated Hospital of Chengdu Medical College, China (Unknown); Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, China (Unknown)
Responsible Party: Principal Investigator, Craig Anderson, Director, Global Brain Health program, The George Institute for Global Health, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTERACT4
Record Dates: First submitted 2018-12-26; First posted 2019-01-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute; Cerebrovascular Disorders
Keywords: stroke; blood pressure control; hypertension; clinical trial; ambulances
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Hypertension | interventions — urapidil

STUDY DESIGN:
Intervention Model Description: central randomization with stratification
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is independent of the treatment team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): If systolic blood pressure>180:IV Urapidil 25mg If systolic blood pressure>150 (or 5 mins after first bolus) : IV Urapidil 25mg and to maintain this level after admission to hospital in those with confirmed acute stroke for the next 7 days (or hospital discharge if earlier)
  Interventions: Drug: urapidil
- control group (No Intervention): To receive blood pressure management according to standard local guidelines which recommend blood pressure lowering in hospital if systolic level is >220mmHg. This level will be considered by ambulance staff as a threshold for treatment if considered clinically important.

INTERVENTIONS:
Drug: urapidil — A standard treatment regime based on intravenous (IV) bolus of 25mg urapidil administered over 1 minute. For those patients initial systolic blood pressure 180, another 25mg urapidil bolus will be given if the systolic blood pressure level persists >150 after 5 minutes.
  Other Names: Intensive BP lowing
  Arms: Intervention group

SUMMARY:
A multicentre, ambulance-delivered, prospective, randomized, open-label, blinded endpoint (PROBE) study to assess the effects of hyperacute intensive blood pressure (BP) lowering initiated in ambulance setting on (i) functional outcome in patients with acute stroke (ii) safety in patients with confirmed acute stroke and other conditions that were initially suspected as acute stroke (i.e. stroke mimic).

DETAILED DESCRIPTION:
As an investigator initiated and conducted, multicentre, ambulance-delivered, prospective, randomised, open-label, blinded outcome (PROBE) study. INTERACT4 aims to evaluate the effects of functional outcome according to an ordinal analysis of the full range of scores on the mRS, the safety in all randomised patients; reperfusion treatment (thrombolysis and/or thrombectomy) related symptomatic ICH (sICH, according to standard definitions), infarct size, the time to and overall rate of reperfusion treatment in AIS patients; hematoma volume and early expansion in ICH.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. Acute syndrome that is due to presumed acute stroke, defined as FAST（Face, Arm, Speech, Time） scores of ≥2 with an arm motor deficit and time ≤2 hours from last seen well;
3. Systolic BP ≥150
4. Able to provide brief informed consent (if a waver of consent is not approved by the ethics committee)

Exclusion Criteria:

1. Coma - no response to tactile stimuli or verbal stimuli;
2. Severe co-morbid disease (e.g. cancer, chronic airflow disease, severe dementia,severe heart failure,pre-stroke disability[needed help]);
3. History of epilepsy or seizure at onset;
4. History of recent head injury (<7 days);
5. Hypoglycemia(glucose<2.8mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2425 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
level of physical function | Day 90
  Level of function defined across 7 categories of disability on the modified Rankin scale （mRS 0-6) in which scores of 0 or 1 indicate good function without or with symptoms but not disability, socress of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.

SECONDARY OUTCOMES:
number of patients with serious adverse events | Day 90
  total number of serious adverse events reported during follow-up, according to standard definitions
number of patients with any intracranial hemorrhage | Day 7
  reperfusion treatment (thrombolysis/thrombectomy) related symptomatic intracerebral number of cases of intracranial hemorrhage, according to standard definitions
size of cerebral infarction | Day 2
  overall size of cerebral infarction on MRI within 2 days in cases of ischaemic stroke
number of patients who receive reperfusion treatment | Day 0
  total number of cases of reperfusion (thrombolysis and/or thrombectomy) in ischemic stroke
time to use of reperfusion treatment | Day 0
  time from symptom onset to reperfusion treatment in patients with ischemic stroke
size of hematoma volume | Day 1
  change in volume of hematoma from baseline to 24 hours, measured on brain imaging
size of hematoma volume | Day 0
  volume of hematoma at baseline measured on brain imaging
death or major disability | Day 90
  Level of function defined across 7 categories of disability on the modified Rankin scale （mRS 0-6) in which scores of 0 or 1 indicate good function without or with symptoms but not disability, socress of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
  mRS(3-6)
Death | Day 90
Disability | Day 90
  Level of function defined across 7 categories of disability on the modified Rankin scale （mRS 0-6) in which scores of 0 or 1 indicate good function without or with symptoms but not disability, socress of 2 indicates slight disability but independence, 3 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
death or dependency measured by a shift in NIHSS | day 1 and day 7
Health related quality of life | day 90
  according to the EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, Principal Investigator — The George Institute for Global Health, China; Lili Song, Principal Investigator — The George Institute for Global Health, China; Gang Li, Principal Investigator — Shanghai East Hospital, China; Jie Yang, Principal Investigator — Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, China; Yapeng Lin, Principal Investigator — The First Affliated Hospital of Chengdu Medical College, China
Locations (4):
- China (4):
  - The George Institute for Global Health, Beijing, Beijing Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, China, Chengdu, Sichuan
  - The First Affliated Hospital of Chengdu Medical College, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with bona fide researchers after 1 year following conclusion of the study, based on a submitted protocol to the research office of The George Institute for Global Health, Sydney Australia
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after conclusion of the study
Access Criteria: genuine researcher with supporting institution protocol review and approval by the research office of The George Institute
URL: http://georgeinstitute.org.au

REFERENCES:
- [Derived] Wang X, Ren X, Li Q, Ouyang M, Chen C, Delcourt C, Chen X, Wang J, Robinson T, Arima H, Ma L, Hu X, You C, Li G, Jie Y, Lin Y, Billot L, Munoz-Venturelli P, Martins S, Pontes-Neto OM, Liu L, Chalmers J, Carcel C, Song L, Anderson CS; INTERACT Investigators. Effects of blood pressure lowering in relation to time in acute intracerebral haemorrhage: a pooled analysis of the four INTERACT trials. Lancet Neurol. 2025 Jul;24(7):571-579. doi: 10.1016/S1474-4422(25)00160-7. PMID 40541207
- [Derived] Li G, Lin Y, Yang J, Anderson CS, Chen C, Liu F, Billot L, Li Q, Chen X, Liu X, Ren X, Zhang C, Xu P, Wu L, Wang F, Qiu D, Jiang M, Peng Y, Li C, Huang Y, Zhao X, Liang J, Wang Y, Wu X, Xu X, Chen G, Huang D, Zhang Y, Zuo L, Ma G, Yang Y, Hao J, Xu X, Xiong X, Tang Y, Guo Y, Yu J, Li S, He S, Mao F, Tan Q, Tan S, Yu N, Xu R, Sun M, Li B, Guo J, Liu L, Liu H, Ouyang M, Si L, Arima H, Bath PM, Ford GA, Robinson T, Sandset EC, Saver JL, Sprigg N, van der Worp HB, Song L; INTERACT4 investigators; INTERACT4 Investigators. Intensive Ambulance-Delivered Blood-Pressure Reduction in Hyperacute Stroke. N Engl J Med. 2024 May 30;390(20):1862-1872. doi: 10.1056/NEJMoa2314741. Epub 2024 May 16. PMID 38752650
- [Derived] Chen C, Lin Y, Liu F, Chen X, Billot L, Li Q, Guo Y, Liu H, Si L, Ouyang M, Zhang C, Arima H, Bath PM, Ford GA, Robinson T, Sandset EC, Saver JL, Sprigg N, van der Worp HB, Liu G, Song L, Yang J, Li G, Anderson CS; INTERACT4 Investigators. Update on the INTEnsive ambulance-delivered blood pressure Reduction in hyper-ACute stroke Trial (INTERACT4): progress and baseline features in 2053 participants. Trials. 2023 Dec 20;24(1):817. doi: 10.1186/s13063-023-07861-5. PMID 38124205
- [Derived] Song L, Chen C, Chen X, Guo Y, Liu F, Lin Y, Billot L, Li Q, Liu H, Si L, Ouyang M, Arima H, Bath PM, Ford GA, Robinson T, Sandset EC, Saver JL, Sprigg N, van der Worp HB, Zhang C, Yang J, Li G, Anderson CS; INTERACT4 investigators. INTEnsive ambulance-delivered blood pressure Reduction in hyper-ACute stroke Trial (INTERACT4): study protocol for a randomized controlled trial. Trials. 2021 Dec 6;22(1):885. doi: 10.1186/s13063-021-05860-y. PMID 34872617